CLINICAL TRIAL: NCT04019379
Title: Calcium and Phosphorus Whole-Body Balance and Kinetics in Patients With Moderate Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1809583731
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Phosphorus and Calcium Disorders; Chronic Kidney Disease Mineral and Bone Disorder; Chronic Kidney Diseases
Keywords: Whole-body balance; Kinetic modeling; Intestinal absorption
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): High Phos crossover to Low Phos
  Interventions: Other: High Phosphorus Diet; Other: Low Phosphorus Diet
- Sequence B (Experimental): Low Phos crossover to High Phos
  Interventions: Other: High Phosphorus Diet; Other: Low Phosphorus Diet

INTERVENTIONS:
Other: High Phosphorus Diet — Controlled research diet of high phosphorus (with low calcium)
Other: Low Phosphorus Diet — Controlled research diet of low phosphorus (with low calcium)

SUMMARY:
This pilot study aims to develop a method for simultaneous whole-body calcium and phosphorus balance and full kinetic modeling of both ions in patients with chronic kidney disease.

DETAILED DESCRIPTION:
The goal of this project is to produce preliminary data on the effects of the commonly prescribed dietary phosphorus restriction on whole-body Calcium (Ca) and Phosphorus (P) balance and kinetics patients with CKD, to support a larger future clinical study. The specific aims are to determine intestinal Ca and P fractional absorption and 2) Ca and P balance and full kinetics, effect sizes variance estimates in patients with CKD on a low Ca diet with high P diet versus dietary P restriction. The hypothesis is that a high P diet, in the context of a typical low Ca diet, leads to P retention negative Ca balance, and that dietary P restriction modestly reduces P retention but does not negative Ca balance.

The study design is a randomized 2-period cross-over study. All outpatient and inpatient visits place at the Indiana CTSI Clinical Research Center located in IU Health University Hospital in Indianapolis, IN. Subjects will be randomly assigned to controlled diets of either low Ca/high P (LCa/HP) or low (LCa/LP) for a 1-week, outpatient diet equilibration period, followed by 1-week inpatient full balance that includes a 48-hour Ca and P absorption testing protocol. After a 1-3 week washout subjects will crossover to the other diet regimen

ELIGIBILITY:
Inclusion Criteria:

* Men or women, ages 30-75 years old, any race or ethnicity
* Moderate chronic kidney disease
* Female subjects must be postmenopausal (>12 months since last menstrual period), surgically sterile, or confirmed not pregnant by pregnancy test
* Must be on stable doses of medications (except those noted in exclusion criteria) for at least 4 weeks prior to the study
* Willing to discontinue nutritional supplements (e.g. vitamin D, calcium, multivitamin/minerals, or others) upon enrollment until completion of the study
* Adequate vitamin D status defined as serum 25D > 20 ng/mL

Exclusion Criteria:

* Plans to initiate dialysis within 6 months
* Hypercalcemia defined as serum calcium >10.5 mg/dL within past 3 months
* Hyperkalemia defined as serum potassium >5.5 mg/dL within past 3 months
* Hyperphosphatemia defined as serum phosphate >5.5 mg/dL within past 3 months
* Intestinal disease that alters absorption or normal intestinal function including celiac disease, small bowel resection, or bariatric surgery
* Serious, uncontrolled underlying systemic disease including diabetes, lupus, hypertension
* Pregnant or breastfeeding
* Prescribed a phosphate binder medication, calcitriol, vitamin D analogs, calcimimetics, parathyroid hormone analogues, and other medications that may alter Ca and P metabolism within past 30 days

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Hill Gallant, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Indiana CTSI CRC, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 71 [71 to 71] | 52 [34 to 69] | 58 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
estimated glomerular filtration rate (eGFR) [Mean (Full Range); unit: mL/min/1.73m^2] | 40 [40 to 40] | 35 [29 to 41] | 37 [29 to 41]
body mass index (BMI) [Mean (Full Range); unit: kg/m^2] | 34.7 [34.7 to 34.7] | 20.5 [19.2 to 21.8] | 25.2 [19.2 to 34.7]
Serum phosphorus [Mean (Full Range); unit: mg/dL] | 2.5 [2.5 to 2.5] | 2.7 [2.6 to 2.8] | 2.6 [2.5 to 2.8]
Serum intact fibroblast growth factor-23 (iFGF23) [Mean (Full Range); unit: pg/mL] | 27.6 [27.6 to 27.6] | 78.3 [77.9 to 78.7] | 61.4 [27.6 to 78.7]
Serum 1,25-dihydroxyvitamin D3 (1,25D) [Mean (Full Range); unit: pg/mL] | 46 [46 to 46] | 26 [21 to 30] | 32 [21 to 46]
Serum intact parathyroid hormone (iPTH) [Mean (Full Range); unit: pg/mL] | 85.5 [85.5 to 85.5] | 154.7 [115.1 to 194.4] | 131.7 [85.5 to 194.4]

OUTCOME MEASURES:

1. Primary Outcome: Fractional Calcium Absorption
Description: Determined by kinetic modeling of serum and urine Ca-44 isotope after oral and IV isotope administrations
Time Frame: 48 hours
Measure: Mean (Full Range); unit: fraction of 1.00
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
fraction of 1.00 | 0.30 [0.22 to 0.45] | 0.42 [0.22 to 0.80]

2. Primary Outcome: Fractional Phosphorus Absorption
Description: Determined by kinetic modeling of serum and urine P-33 isotope after oral and IV isotope administrations
Time Frame: 48 hours
Measure: Mean (Full Range); unit: fraction of 1.00
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
fraction of 1.00 | 0.73 [0.58 to 0.95] | 0.69 [0.51 to 0.91]

3. Primary Outcome: Calcium Balance
Description: Determined by analysis of calcium content in complete 24-hour urine and stool collections, subtracted from the diet calcium content consumed. Values can be negative, zero, or positive.
Time Frame: 1 week
Measure: Mean (Full Range); unit: mg/d
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
mg/d | 126 [-36 to 343] | 199 [117 to 315]

4. Primary Outcome: Phosphorus Balance
Description: Determined by analysis of phosphorus content in complete 24-hour urine and stool collections, subtracted from the diet phosphorus content consumed. Values can be negative, zero, or positive.
Time Frame: 1 weeks
Measure: Mean (Full Range); unit: mg/d
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
mg/d | 65 [-292 to 481] | 73 [-144 to 416]

5. Secondary Outcome: Serum Intact Fibroblast Growth Factor 23 (iFGF23)
Description: Determined by enzyme-linked immunoassay (ELISA). Values for each subject are an average of 6 serial measures taken during the 1 week balance period (between Days 1-8)
Time Frame: Day 1-8
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
pg/mL | 67.9 [47.9 to 96.2] | 53.4 [44.1 to 68.6]

6. Secondary Outcome: Serum Intact Parathyroid Hormone (iPTH)
Description: as for outcome 5
Time Frame: Day 1-8
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
pg/mL | 122.7 [101.2 to 136.2] | 104.7 [92.2 to 113.4]

7. Secondary Outcome: Serum 1,25-dihydroxyvitamin D (1,25D)
Description: Determined by LC-MS/MS. Values are from Day 1 of the metabolic balance period (following 1 week of acclimation to assigned study diet).
Time Frame: Day 1
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
Number analyzed (Participants) | 3 | 3
pg/mL | 29.7 [21 to 40] | 29.7 [17 to 41]

ADVERSE EVENTS:
Time Frame: Time of enrollment through study completion, approximately 2 months.
Arm/Group | High Phosphorus Diet | Low Phosphorus Diet
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT04019379/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT04019379/ICF_001.pdf